CLINICAL TRIAL: NCT04992884
Title: Body Surface Gastric Mapping to Evaluate Patients With Upper Gastrointestinal Symptoms and Controls
Brief Title: Non-invasive Measurement of Gastric Motility
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Greg O'Grady (Other)
Responsible Party: Sponsor-Investigator, Greg O'Grady, Professor, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Other Study IDs: CLD-014
Record Dates: First submitted 2021-07-14; First posted 2021-08-05 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Adults,Gastric Symptoms,Suspected Gastric Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Gastric Alimetry — Gastric Alimetry is a medical device intended to record, store, view and process gastric myoelectrical activity as an aid in the diagnosis of gastrointestinal motility disorders. The device is indicated for use during the diagnostic work-up of patients reporting gastric symptoms, who are suspected of having an underlying gastric motility problem.
  Other Names: Medtronic Polygram NET / Polygraf ID EGG system

SUMMARY:
Clinical evaluation to compare performance of the physiological recordings from the Gastric Alimetry System vs a predicate reference device (Medtronic Polygram NET / Polygraf ID EGG System

DETAILED DESCRIPTION:
A prospective, non-randomised, single centre investigation on patients with suspected motility disorders comprising a simultaneous head-to-head comparison of device performance between the Gastric Alimetry System and the Medtronic Polygram NET / Polygraf ID EGG System.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 years old or older
* Able to provide written informed consent
* Patients with a suspected motility disorder, meetingRome IVCriteria for functional dyspepsia or chronic nausea and vomiting syndromes or having a diagnosis of gastroparesis as confirmed by a standardized gastric scintigraphy study, including having >10% gastric meal retention at 4-hours.

Exclusion Criteria:

* BMI >35 kg m(2)
* Known metabolic, neurogenic or endocrine disorders known to cause gastrointestinal dysmotility e.g. multiple sclerosis, Parkinson's disease, hypothyroidism
* Known current gastrointestinal infection (includes H.pylori when being actively treated)
* Known current inflammatory bowel disease
* Known current gastrointestinal malignancy
* Previous gastroduodenal surgery
* Open abdominal wounds or abdominal skin not intact (e.g.rash, abrasions, weeping tissues)
* Fragile skin evidenced by high susceptibility to skin tears or skin that bruises easily
* Regular cannabis use
* Allergy to adhesives
* Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adult patients with upper gastrointestinal symptoms suspected to have gastric motility disorders.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Performance comparison (frequency) between Gastric Alimetry and predicate device | 90 minutes
  Mean frequency of raw data from predicate device compared with the same measure from the Gastric Alimetry System. Electrode placement is identical and recording is simultaneous.

SECONDARY OUTCOMES:
Performance comparison (amplitude) between Gastric Alimetry and predicate device | 90 minutes
  Mean amplitude of raw data from predicate device (4 electrodes) compared with the same measure from the Gastric Alimetry System (4 electrodes). Electrode placement is identical and recording is simultaneous.
Performance comparison (amplitude) between Gastric Alimetry (4 channels as per Primary Outcome Measure) and Gastric Alimetry (8 highest amplitude electrodes). | 90 minutes
  Amplitude of raw data from Gastric Alimetry device (4 electrodes) compared with the same measure from the Gastric Alimetry System (8 electrodes with highest amplitude). Recording is simultaneous.
Safety Endpoint | Five hours
  Safety endpoint: no unanticipated AEs or ADEs, and anticipated AEs and ADEs are acceptable relative to the risk acceptability criteria, as defined by the risk acceptability matrix (RSK-010).
User Needs Endpoint | Five hours
  User needs validation results meet acceptability criteria.

CONTACTS AND LOCATIONS:
Overall Officials: John A Windsor, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Clinical Research Centre, Building 507, The University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided